CLINICAL TRIAL: NCT05098873
Title: Study on High Potential in Adolescence School Boredom as a Precursor to a Depressive Episode Single-center, Comparative Study of High School Students
Brief Title: Study on Boredom in High Potential Adolescents
Acronym: ESchAHP
Status: Completed | Type: Observational
Sponsor: Centre Psychothérapique de Nancy (Other)
Responsible Party: Sponsor
Other Study IDs: RIPH 2021-02; 2021-A01118-33 (Other: ANSM (French competent authority))
Record Dates: First submitted 2021-10-20; First posted 2021-10-28 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Intelligence; Boredom
Keywords: Intelligence; Boredom

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group gifted teens
  Interventions: Other: psychodynamic
- Group no gifted teens
  Interventions: Other: psychodynamic

INTERVENTIONS:
Other: psychodynamic — intervention with adolescents through the presentation of questions to be completed

SUMMARY:
The research focuses on "High Potential" (HP) in adolescence, in a link with the professional practice of the investigators.

Furthermore, supported by scientific literature and professional clinical practice, this research is interested in school boredom, regularly expressed by the consulting adolescents, in its relation with a depressive syndrome.

The objective of the research is to know if school boredom is a precursor of a depressive episode in high school students with HP compared to high school students without HP.

DETAILED DESCRIPTION:
The investigators are questioning the meaning of school boredom experienced by adolescents with HP and its link with a depressive syndrome. The investigators will use clinical interviews, rating scales for a quantitative measure and projective tests for a psychodynamic study. The responses of adolescents with HP will be compared to those of adolescents without HP.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents coming for consultation in a medical-psychological center of Sponsor
* Adolescents aged 14 to 16 years and 11 months.
* Adolescents expressing a psychological malaise and/or an anxiety disorder at the time of the consultation request
* Adolescents who were informed about the study, received the information note about it and did not object to participating
* At least one parent or guardian who was informed of the study, received the study information sheet, and did not object to the child's participation
* Adolescents affiliated or entitled to a social security plan

Exclusion Criteria:

* Adolescents who do not understand the French language well enough to complete the questionnaires.
* Adolescents with a clear diagnosis of psychiatric pathology (e.g. schizophrenia)
* Adolescents with an IQ ≤ 80 because the level of intellectual efficiency would be too fragile and too far from the expectations of our research.

Ages: 14 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Adolescents consulting the medical-psychological centers of our hospital (Centre Psychothérapique de Nancy = Sponsor) for psychological malaise and/or anxiety-depressive disorders and academic difficulties
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
Wechsler Intelligence Scale for Children | Month 2 or 3
  Intelligence test that measures a child's intellectual ability and 5 cognitive domains that impact performance.
Échelle de Disposition à l'Ennui (French Title) | Month 1 or 2
  Boredom scale It is the French adaptation of the Boredom Proneness Scale
Rorschach test | Month 3
  Projective test
Thematic Apperception Test | Month 3
  Projective test

SECONDARY OUTCOMES:
Multidimensional Anxiety Scale for Children | Month 1 or 2
  Anxiety scale
Children Depression Inventory | Month 1 or 2
  Depression scale
Self-Perception Profile for Adolescents | Month 1 or 2
  Self-esteem scale This self-report scale taps how adolescents assess their "competence" or "adequacy" in different areas of their life, and how they evaluate their overall self-worth as a person.

CONTACTS AND LOCATIONS:
Overall Officials: Valérie BURGÉ, Principal Investigator — Centre Psychothérapique de Nancy
Locations (1):
- Centre Psychothérapique de Nancy - CMP Adolescents Lunéville, Lunéville, France

IPD SHARING:
Plan to Share IPD: No